CLINICAL TRIAL: NCT05550376
Title: Genotype-phenotype Association Study of ENG and ACVRL1 Genes in the Inflammatory and Endothelial Response in Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Genotype-phenotype Association in Hereditary Hemorrhagic Telangiectasia
Acronym: Generate-HHT
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Sociedad Española De Medicina Interna (Other)
Responsible Party: Sponsor
Other Study IDs: 301/20
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; HHT; Rendu Osler Weber Disease
Keywords: Hereditary Hemorrhagic Telangiectasia; HHT; Rendu Osler Weber Disease; Genotype-phenotype association; ENG; ALK-1
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Plasma (EDTA and citrate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HHT1: Mutations in the ENG (endoglin) gene
  Interventions: Other: Registry
- HHT2: Mutations in the ALK-1 (activin receptor-like kinase) gene
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Non-interventional registry

SUMMARY:
The present project aims to study the inflammatory and endothelial responses involved in the differences in clinical events related to both genotypes (ENG vs. ACVRL1) in HHT. Accordingly, a cross-sectional study is proposed to evaluate the differences in circulating inflammatory and endothelial biomarkers, including interleukines, adhesion molecules, chemokines and immune regulatory molecules between both HHT groups.

DETAILED DESCRIPTION:
Background and rationale: Hereditary Hemorrhagic Telangiectasia (HHT) is a rare disease characterized by a multisystemic vascular dysplasia with autosomal dominant inheritance, mainly caused by mutations in ENG and ACVRL1 genes. Even though those mutations have been related to different clinical manifestations, the molecular mechanisms involved in each genetic variant have not been clarified. Methods: A cohort study will be carried out to compare the incidence of clinical events after a 12-months follow-up. The ability of these biomarkers to predict the clinical events will be assessed in a multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Confirmed diagnosis of HHT, according to the Curaçao criteria or genetic diagnosis.
* Clinically stable condition at the time of inclusion, defined as score < 7 points on the Epistaxis Severity Score (ESS).
* Having signed the informed consent, after having received all the information concerning the study.

Exclusion Criteria:

* Major coronary or cerebrovascular event in the 3 months prior to inclusion.
* Serious intercurrent illnesses, such as acute infections, outbreaks of autoimmune or inflammatory pathology, active cancer, or other pathologies that, at the investigator's discretion, could interfere with the conduct of the study.
* Major surgery during the 2 months prior to inclusion.
* Pharmacological treatment maintained during the 3 months prior to inclusion with NSAIDs, corticosteroids or chemotherapy.
* Toxic habits, including severe smoking, alcohol or drug abuse, which in the opinion of the investigator could interfere with the conduct of the study.
* Pregnancy or puerperium.
* Any other condition that limits compliance with the visits or procedures established in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive sample of patients with HHT will be selected from the subjects under follow-up in the Internal Medicine Department of the Hospital Universitario Ramón y Cajal.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hemorrhagic clinical events | 12-month follow-up period after inclusion
  Presence of significant bleeding of any location, recurrent and/or massive, or performance of therapeutic procedures to control them.

SECONDARY OUTCOMES:
Other significant clinical events | 12-month follow-up period after inclusion
  Significant clinical events other than hemorrhagic episodes (e.g., infections, neoplasms or other severe diseases)
Changes in quality of life | 12-month follow-up period after inclusion
  Significant changes in quality of life as measured by the EuroQol 5-level EQ-5D version (EQ-5D-5L) and the EuroQol visual analogue scale (EQ VAS).
  EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The index ranges from 1 (best state of health) to 0 (death).
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100 points) and 'The worst health you can imagine' (0 points).

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Patier, MD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Viteri-Noel A, Gonzalez-Garcia A, Patier JL, Fabregate M, Bara-Ledesma N, Lopez-Rodriguez M, Gomez Del Olmo V, Manzano L. Hereditary Hemorrhagic Telangiectasia: Genetics, Pathophysiology, Diagnosis, and Management. J Clin Med. 2022 Sep 5;11(17):5245. doi: 10.3390/jcm11175245. PMID 36079173
- [Background] Sanchez-Martinez R, Iriarte A, Mora-Lujan JM, Patier JL, Lopez-Wolf D, Ojeda A, Torralba MA, Juyol MC, Gil R, Anon S, Salazar-Mendiguchia J, Riera-Mestre A; RiHHTa Investigators of the Rare Diseases Working Group from the Spanish Society of Internal Medicine. Current HHT genetic overview in Spain and its phenotypic correlation: data from RiHHTa registry. Orphanet J Rare Dis. 2020 Jun 5;15(1):138. doi: 10.1186/s13023-020-01422-8. PMID 32503579
- [Background] Albinana V, Gimenez-Gallego G, Garcia-Mato A, Palacios P, Recio-Poveda L, Cuesta AM, Patier JL, Botella LM. Topically Applied Etamsylate: A New Orphan Drug for HHT-Derived Epistaxis (Antiangiogenesis through FGF Pathway Inhibition). TH Open. 2019 Jul 26;3(3):e230-e243. doi: 10.1055/s-0039-1693710. eCollection 2019 Jul. PMID 31360828
- See also: The Multisystemic Diseases Group encompasses several lines of research related to pathologies that involve complex clinical management that usually falls within the scope of Internal Medicine. — http://www.irycis.org/en/research/research-groups/43/multisystemic-diseases